CLINICAL TRIAL: NCT05753228
Title: In Vivo Investigation on Mitochondrial Dysfunction in Post-COVID Fatigue and Cancer Fatigue.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DSRB 2022/00668
Record Dates: First submitted 2023-03-02; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-01

CONDITIONS: Mitochondrial Dysfunction; COVID-19; Fatigue
Keywords: Mitochondrial dysfunction; COVID-19 fatigue; Cancer fatigue
MeSH Terms: conditions — Mitochondrial Diseases; COVID-19; Fatigue | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Case-control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID fatigue patients (Active Comparator): MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS),Chalder fatigue scale, Health Questionnaire (EQ-5D-5L), Hamilton Depression Rating Scale
  Interventions: Other: MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS); Other: Chalder Fatigue Scale; Other: Health Questionnaire (EQ-5D-5L); Other: Hamilton Depression Rating Scale
- Cancer fatigue patients (Active Comparator): MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS),Chalder fatigue scale, Health Questionnaire (EQ-5D-5L), Hamilton Depression Rating Scale
  Interventions: Other: MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS); Other: Chalder Fatigue Scale; Other: Health Questionnaire (EQ-5D-5L); Other: Hamilton Depression Rating Scale
- Healthy patients as controls (Active Comparator): MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS),Chalder fatigue scale, Health Questionnaire (EQ-5D-5L), Hamilton Depression Rating Scale
  Interventions: Other: MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS); Other: Chalder Fatigue Scale; Other: Health Questionnaire (EQ-5D-5L); Other: Hamilton Depression Rating Scale

INTERVENTIONS:
Other: MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) — MRI/ 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) to assess metabolic and mitochondrial perturbations in post-COVID fatigue or cancer fatigue.
Other: Chalder Fatigue Scale — The Chalder Fatigue Scale is used for measuring the extent and severity of fatigue within both clinical and non-clinical, epidemiological populations.
Other: Health Questionnaire (EQ-5D-5L) — The Health Questionnaire (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."
Other: Hamilton Depression Rating Scale — The Hamilton Depression Rating Scale is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.

SUMMARY:
To date, little is understood regarding post-COVID fatigue or cancer fatigue though it is known to affect a large proportion of patients (10-70% depending on the population). This study aims to investigate potential mitochondrial function and metabolic changes in brain to provide further information regarding the etiology of these changes leading to fatigue.

This study hypothesized that Post-COVID fatigue is ensued by perturbations in metabolism and mitochondrial function in the brain.

This is a case-control study. In this study, 30 patients (experimental group) complaining of persistent fatigue lasting longer than 4 weeks after recovering from SARS-CoV-2 infection and the age/gender-matched control of 30 healthy subjects (control group 1) and 30 patients suffering from cancer-related fatigue patients longer than 4 weeks after remission (control group 2). Both the experimental group (post-COVID fatigue) and control group 2 (cancer fatigue) will be recruited from NUH outpatient clinic will undergo a session of MRI, 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) and the Chalder Fatigue Scale, Health Questionnaire (EQ-5D-5L) and Hamilton Depression Rating Scale at baseline and follow-up visit.

DETAILED DESCRIPTION:
The clinical manifestations of post-COVID fatigue are comparable with chronic fatigue syndrome or myalgic encephalomyelitis (CFS/ME) whose clinical features comprise substantial decrease in function persisting for more than 6 months, post-exertional malaise, unrefreshing sleep, cognitive impairment or orthostatic intolerance (Blomberg, 2021; Logue, 2021). From the clinical perspective, there is high plausibility of abnormalities of energy production or mitochondrial function as the etiology of CFS/ME (Tomas, 2017; Filler, 2014). The similar clinical features were observed in other infections such as EBV, Ebola, lime disease, etc., which led to coining a terminology, post-infectious syndrome. Considering the recent study showing SARS-CoV-2 reduces mitochondrial proteins uniquely, known as Complex One, to quiet the cell's metabolic output (Miller, 2021), the etiological relevance of post-COVID fatigue and CFS/ME should be scrutinized. By the way, fatigue is prevalent in cancer survivors even after achieving the complete remission, which is described as "paralyzing" and ensues physical or mental exhaustion that may not reversed by taking rest or sleep. This cancer related fatigue may compound the effect of chemo brain or chemo fog which denotes cancer-related cognitive dysfunction lingering for months or years after cancer treatment. As such, there are many analogous clinical features shared by post-COVID fatigue and cancer fatigue. The comparison of the metabolic changes between post-COVID fatigue and cancer fatigue may provide hints to understand the mechanism of fatigue better.

It has been challenging technically to verify the role of mitochondria in CFS/ME. A commercially available test, e mitochondrial energy score protocol, failed to show the reliability and reproducibility required of a diagnostic test (Thomas, 2019), which implies the practical limitations of in vitro test to evaluate mitochondrial function given the intrinsic and extrinsic factors affecting the test result of target metabolites. That said, proton Magnetic Resonance spectroscopy (MRS) can be a useful tool which detects the major brain metabolites such as N-acetylaspartate (NAA), creatinine (Cr), myo-inositol (MI) and lactate (Kantarci, 2003). The MRS spectra including abnormal positive lactate peaks correlate well with other clinical markers in mitochondriopathies (Lin, 2003). The level of organic acid (including 3-methylglutacoric acid) in urine is associated with compromised mitochondrial energy metabolism (Ikon N, 2016), which will be used as an adjunct index.

To date, little is understood regarding post-COVID fatigue or cancer fatigue though it is known to affect a large proportion of patients (10-70% depending on the population). This study aims to investigate potential mitochondrial function and metabolic changes in brain to provide further information regarding the etiology of these changes leading to fatigue.

This study aims:

1) to determine whether there are changes in the NAA/MI indicating perturbed bioenergetic role in neuronal mitochondrial function in post-COVID fatigue and 2) to prove changes of cerebral blood flow (CBF) assessed by 3D Arterial Spin Labelling (ASL) sequence for brain in post-COVID fatigue.

This study hypothesized that Post-COVID fatigue is ensued by perturbations in metabolism and mitochondrial function in the brain.

This study will include 30 patients (experimental group) complaining of persistent fatigue lasting longer than 4 weeks after recovering from SARS-CoV-2 infection and the age/gender-matched control of 30 healthy subjects (control group 1) and 30 patients suffering from cancer-related fatigue patients longer than 4 weeks after remission (control group 2). Both the experimental group (post-COVID fatigue) and control group 2 (cancer fatigue) will be recruited from NUH outpatient clinic. The healthy control will be recruited from NUH employees from various work groups utilizing a recruitment flyer and word of mouth.

Screening Visits and Procedures:

(Visit 1) The study details will be explained clearly to the prospective participants and consent will be taken from the participants prior to commencing study procedures which includes screening, accessing and extracting data from their medical records, administering the study questionnaires (Chalder fatigue scale) and arranging for the study participants to undergo MRI, 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) at the NUS-Center for transitional magnetic resonance (TMR). Eligible subjects will then proceed to the following visits.

Visit 2 which will take place within 28 days of the first visit and will involve MRI/MRS/ASL measurements to assess metabolic and mitochondrial perturbations in post-COVID fatigue or cancer fatigue (details below). The urine sample (10ml) will be collected from all subjects to measure changes of organic acid level against normal range which may reflect mitochondrial dysfunction.

Final Study Visit (3rd visit or phone call). For the participants in the post-COVID fatigue group and the cancer fatigue group, the study team will apply the same questionnaires including Chalder Fatigue Scale, Health Questionnaire (EQ-5D-5L) and Hamilton Depression Rating Scale through a phone call or in person, which will coincide with their follow up visit with their treating physician. For healthy normal subjects without fatigue symptoms, the questionnaires will be administered via a phone call and do not need to attend Visit 3 in person, which is set to monitor the clinical course of post-COVID fatigue and cancer fatigue.

This is a case-control study. With a sample size of 30 per group (90 in total for 3 groups), the study will have 90% power to detect a standard difference of 0.95 and the mean difference in the primary endpoints equal to 95% of the SD of the endpoint. As such, the minimum sample size will be at least 27 per group. Since the two primary endpoints of the study are NAA/MI measured by proton MRS and cerebral blood flow (CBF) assessed by 3D Arterial Spin Labelling (ASL) sequence for brain, the significant level will be adjusted to 0.0125 (for 2 primary endpoints and 2 controls, the significant level will be 0.05/4).

Those numerical variables measured in MRI/MRS will be compared with either healthy control or disease control (cancer fatigue patients). 2 sample T test or Mann-Whitney U test, whichever is more appropriate for the hypothesis testing will be used. Linear regression can be applied to adjust for other confounders or covariates.

The Null hypothesis: the mean NAA/MI and CBF of study group equals to the mean NAA/MI and CBF of disease control group (cancer fatigue) and healthy control group. The alternative hypothesis: the mean NAA/MI and CBF of study group is different from the mean NAA/MI and CBF of disease control group and healthy control group.

Type I error: 0.0125 Type II error: 0.1

ELIGIBILITY:
Inclusion Criteria:

* age between 21 and 70 years old (all 3 groups)
* SARS-COV-2 disease confirmed by PCR or ART (experimental group)
* Chalder Fatigue Score (CFQ-11): >= 19 (experimental group and control group 2), =< 11 (control group 1)
* able to understand the study purpose and consent to it (all 3 groups)

Exclusion Criteria:

* medically unstable
* contraindications for MR scanning (metallic implants, claustrophobia)
* requiring oxygen supplementation
* unable to follow instructions
* anemia (Hb < 10g/dl)
* thyroid disorder
* neoplasm (applicable only to experimental group and control group 1)
* premorbid sleep disorder
* premorbid psychiatric disorders including depression
* pregnancy
* epilepsy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2023-12-08 (Estimated)

PRIMARY OUTCOMES:
MRI, 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) | 90 minutes
  The MRI, 3D Arterial Spin Labelling (ASL) and 1H magnetic resonance spectroscopy (MRS) are used to assess metabolic and mitochondrial perturbations in post-COVID fatigue or cancer fatigue.
Chalder Fatigue Scale | 5 minutes
  Chalder Fatigue Scale is a self-administered questionnaire for measuring the extent and severity of fatigue within both clinical and non-clinical, epidemiological populations. Each of the 11 items are answered on a 4-point scale ranging from the asymptomatic to maximum symptomology, such as 'Better than usual', 'No worse than usual', 'Worse than usual' and 'Much worse than usual'. For all items, the least symptomatic answers are on the left of the response-set, providing an easy-to-understand checklist for respondents. Using the Likert scoring method, responses on the extreme left receive a score of 0, increasing to 1, 2 or 3 as they become more symptomatic. The respondent's global score can range from 0 to 33. The global score also spans two dimensions-physical fatigue (measured by items 1-7) and psychological fatigue (measured by items 8-11). The Likert scoring system allows for means and distributions to be calculated for both the global total as well as the two sub-scales.
Health Questionnaire (EQ-5D-5L) | 5 minutes
  The Health Questionnaire (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems." The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Hamilton Depression Rating Scale | 10 minutes
  The Hamilton Depression Rating Scale is used to quantify the severity of symptoms of depression and is one of the most widely used and accepted instruments for assessing depression. Method for scoring varies by version. For the HDRS17, a score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher (indicating at least moderate severity) is usually required for entry into a clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon K Lim, MD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Jeong Hoon K Lim, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared to other researchers.

REFERENCES:
- [Background] Blomberg B, Mohn KG, Brokstad KA, Zhou F, Linchausen DW, Hansen BA, Lartey S, Onyango TB, Kuwelker K, Saevik M, Bartsch H, Tondel C, Kittang BR; Bergen COVID-19 Research Group; Cox RJ, Langeland N. Long COVID in a prospective cohort of home-isolated patients. Nat Med. 2021 Sep;27(9):1607-1613. doi: 10.1038/s41591-021-01433-3. Epub 2021 Jun 23. PMID 34163090
- [Background] Filler K, Lyon D, Bennett J, McCain N, Elswick R, Lukkahatai N, Saligan LN. Association of Mitochondrial Dysfunction and Fatigue: A Review of the Literature. BBA Clin. 2014 Jun 1;1:12-23. doi: 10.1016/j.bbacli.2014.04.001. PMID 25147756
- [Background] Logue JK, Franko NM, McCulloch DJ, McDonald D, Magedson A, Wolf CR, Chu HY. Sequelae in Adults at 6 Months After COVID-19 Infection. JAMA Netw Open. 2021 Feb 1;4(2):e210830. doi: 10.1001/jamanetworkopen.2021.0830. PMID 33606031
- [Background] Miller B, Silverstein A, Flores M, Cao K, Kumagai H, Mehta HH, Yen K, Kim SJ, Cohen P. Host mitochondrial transcriptome response to SARS-CoV-2 in multiple cell models and clinical samples. Sci Rep. 2021 Jan 8;11(1):3. doi: 10.1038/s41598-020-79552-z. PMID 33420163
- [Background] Tomas C, Brown A, Strassheim V, Elson JL, Newton J, Manning P. Correction: Cellular bioenergetics is impaired in patients with chronic fatigue syndrome. PLoS One. 2018 Feb 8;13(2):e0192817. doi: 10.1371/journal.pone.0192817. eCollection 2018. PMID 29420633
- [Background] Tomas C, Lodge TA, Potter M, Elson JL, Newton JL, Morten KJ. Assessing cellular energy dysfunction in CFS/ME using a commercially available laboratory test. Sci Rep. 2019 Aug 7;9(1):11464. doi: 10.1038/s41598-019-47966-z. PMID 31391529
- [Background] Kantarci K, Reynolds G, Petersen RC, Boeve BF, Knopman DS, Edland SD, Smith GE, Ivnik RJ, Tangalos EG, Jack CR Jr. Proton MR spectroscopy in mild cognitive impairment and Alzheimer disease: comparison of 1.5 and 3 T. AJNR Am J Neuroradiol. 2003 May;24(5):843-9. PMID 12748083
- [Background] Lin DD, Crawford TO, Barker PB. Proton MR spectroscopy in the diagnostic evaluation of suspected mitochondrial disease. AJNR Am J Neuroradiol. 2003 Jan;24(1):33-41. PMID 12533324